CLINICAL TRIAL: NCT06730451
Title: Washed Microbiota Transplantation for Postoperative Complications in Solid Organ Transplantation
Brief Title: Microbiota Transplantation in Solid Organ Transplantation
Status: Recruiting | Type: Observational
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: The Chinese fmtBank (Unknown)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Other Study IDs: WMT-SOT complications
Record Dates: First submitted 2024-12-06; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Solid Organ Transplant Complications
Keywords: Solid Organ Transplant Complications; Washed microbiota transplantation; Fecal microbiota transplantation; Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fecal, urine, and blood samples before and after intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Washed Microbiota Transplantation — Washed microbiota suspension delivered through mild-gut and lower-gut

SUMMARY:
Solid organ transplantation (SOT), an alternative therapy for end-stage diseases, offers increased longevity and better quantity of life. Posttransplant complications such as gastrointestinal symptoms, infection, and graft rejection increase risk with graft failure and death. However, the treatment of abovementioned complications remains unsatisfactory. Gut dysbiosis has been reported in patients with SOT, especially in patients with posttransplant complications. Recipients are more susceptible to gut dysbiosis as long-term use of immunosuppressants, antibiotics and corticosteroids. Restoring gut microbiome may be a promising therapy for posttransplant complications. Washed microbiota transplantation (WMT) is a newly improved methodology of fecal microbiota transplantation based on automatic facilities, washing process and a new delivery routine. In this study, investigators aimed to evaluate the efficacy and safety of WMT for postoperative complications in SOT.

ELIGIBILITY:
Inclusion Criteria:

1. solid organ transplantation recipients;
2. suffering from gastrointestinal symptoms (e.g. diarrhea, constipation, abdominal pian), infection (e.g. Clostridium difficile) post-transplantation and so on;
3. is willing to undergo WMT and provide written informed consent.

Exclusion Criteria:

1. patients with history of gastrointestinal diseases or homologous pathogen infection pre-transplant;
2. pregnant or lactating females;
3. expected survival<1 months;
4. unable to understand the purpose of the study, communicate effectively with investigators and comply with all study procedures;
5. follow up less than 1-month post-WMT;
6. other conditions judged by investigators not suitable for study participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Solid organ transplantation recipients receiving WMT will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Stool frequency and consistency | Baseline, 1-week, 2-week, 1-month, 2-month, 3-month post WMT
  Stool frequency ≥3 times per day was considered as diarrhea. Higher frequency represents more severe diarrhea. Stool consistency will be evaluated according to the Bristol Stool Form Scale ranging from type 1 - type 7. Type 1 and 2 indicate constipation, Type 3 and type 4 indicate normal defecation, Type 5, 6 and 7 indicate diarrhea.
Gastrointestinal Symptom Rating Scale (GSRS) | Baseline, 1-week, 2-week, 1-month, 2-month, 3-month post WMT
  GSRS is a 15-item instrument designed to assess the symptoms associated with common GI disorders. The GSRS consists of 5 subscales (reflux, diarrhea, constipation, abdominal pain, and indigestion) producing a mean subscale score ranging from 1 (no discomfort) to 7 (very severe discomfort).

SECONDARY OUTCOMES:
The changes in gut microbiota composition by sequencing faecal metagenome | Baseline, 1-month, 3-month post WMT
  The changes in gut microbe composition before and after WMT were evaluated by sequencing faecal metagenome.
Quality of life by 36-Item Short Form Health Survey(SF-36) | Baseline, 1-month, 3-month post WMT
  SF-36 is a 36-item questionnaire to assess the impact of disease on daily life. The SF-36 consists of 8 subscales (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health) ranging from 0 to 100. Lower scores represent more dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gabarre P, Loens C, Tamzali Y, Barrou B, Jaisser F, Tourret J. Immunosuppressive therapy after solid organ transplantation and the gut microbiota: Bidirectional interactions with clinical consequences. Am J Transplant. 2022 Apr;22(4):1014-1030. doi: 10.1111/ajt.16836. Epub 2021 Oct 15. PMID 34510717
- [Background] Lee JR, Magruder M, Zhang L, Westblade LF, Satlin MJ, Robertson A, Edusei E, Crawford C, Ling L, Taur Y, Schluter J, Lubetzky M, Dadhania D, Pamer E, Suthanthiran M. Gut microbiota dysbiosis and diarrhea in kidney transplant recipients. Am J Transplant. 2019 Feb;19(2):488-500. doi: 10.1111/ajt.14974. Epub 2018 Jul 21. PMID 29920927
- [Background] Swarte JC, Li Y, Hu S, Bjork JR, Gacesa R, Vich Vila A, Douwes RM, Collij V, Kurilshikov A, Post A, Klaassen MAY, Eisenga MF, Gomes-Neto AW, Kremer D, Jansen BH, Knobbe TJ, Berger SP, Sanders JF, Heiner-Fokkema MR, Porte RJ, Cuperus FJC, de Meijer VE, Wijmenga C, Festen EAM, Zhernakova A, Fu J, Harmsen HJM, Blokzijl H, Bakker SJL, Weersma RK. Gut microbiome dysbiosis is associated with increased mortality after solid organ transplantation. Sci Transl Med. 2022 Aug 31;14(660):eabn7566. doi: 10.1126/scitranslmed.abn7566. Epub 2022 Aug 31. PMID 36044594
- [Background] Cheng YW, Phelps E, Ganapini V, Khan N, Ouyang F, Xu H, Khanna S, Tariq R, Friedman-Moraco RJ, Woodworth MH, Dhere T, Kraft CS, Kao D, Smith J, Le L, El-Nachef N, Kaur N, Kowsika S, Ehrlich A, Smith M, Safdar N, Misch EA, Allegretti JR, Flynn A, Kassam Z, Sharfuddin A, Vuppalanchi R, Fischer M. Fecal microbiota transplantation for the treatment of recurrent and severe Clostridium difficile infection in solid organ transplant recipients: A multicenter experience. Am J Transplant. 2019 Feb;19(2):501-511. doi: 10.1111/ajt.15058. Epub 2018 Aug 31. PMID 30085388
- [Background] Swarte JC, Douwes RM, Hu S, Vich Vila A, Eisenga MF, van Londen M, Gomes-Neto AW, Weersma RK, Harmsen HJM, Bakker SJL. Characteristics and Dysbiosis of the Gut Microbiome in Renal Transplant Recipients. J Clin Med. 2020 Feb 1;9(2):386. doi: 10.3390/jcm9020386. PMID 32024079
- [Background] Zhang T, Lu G, Zhao Z, Liu Y, Shen Q, Li P, Chen Y, Yin H, Wang H, Marcella C, Cui B, Cheng L, Ji G, Zhang F. Washed microbiota transplantation vs. manual fecal microbiota transplantation: clinical findings, animal studies and in vitro screening. Protein Cell. 2020 Apr;11(4):251-266. doi: 10.1007/s13238-019-00684-8. Epub 2020 Jan 9. PMID 31919742
- [Background] Lu G, Wang W, Li P, Wen Q, Cui B, Zhang F. Washed preparation of faecal microbiota changes the transplantation related safety, quantitative method and delivery. Microb Biotechnol. 2022 Sep;15(9):2439-2449. doi: 10.1111/1751-7915.14074. Epub 2022 May 16. PMID 35576458